CLINICAL TRIAL: NCT04219852
Title: Contraception and Bariatric Surgery: Evaluation of Contraception and Contraceptive Knowledge of Women Undergoing Bariatric Surgery at the University Hospital of Reims
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO19121*
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Bariatric Surgery Candidate
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- "bariatric surgery" group: Women between 18 and 50 years, who undergone bariatric surgery at the University Hospital of Reims.
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — data collection

SUMMARY:
Obesity is a public health phenomenon affecting more than 17% of women in France, and more than 20% of men and women in Champagne-Ardenne.

Obese women are more likely to have an unplanned pregnancy, whereas these pregnancies are more at risk than women of normal weight and should be planned or considered after weight loss. These women are also often less well followed in terms of gynecology and especially on contraception.

More and more patients are opting for bariatric surgery. However, bariatric surgery is not trivial. Indeed, the important loss of weight expected is at risk of nutritional deficiencies. In addition, a large number of patients are still obese during the months following surgery. This is why pregnancy is theoretically contraindicated within 12 or 18 months postoperatively.

Women with bariatric surgery must have been properly informed of these risks so that they can choose a contraceptive method, and that can be adapted to both their risk factors and the surgical technique performed.

DETAILED DESCRIPTION:
The purpose of this study is to describe contraception in obese women who have undergone bariatric surgery in Champagne-Ardenne.

ELIGIBILITY:
Inclusion Criteria:

* Women between 18 and 50 years old
* Followed at Reims University Hospital after bariatric surgery
* Pre-menopausal status
* Accepting to participate in the study

Exclusion Criteria:

* Women less than 18 or more than 50 years old
* Women with postmenopausal status
* Women refusing to participate

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women between 18 and 50 years, pre-menopausal, who undergone bariatric surgery at Reims University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2020-04-14 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
contraception method | Day 0
  Presence of contraception during the postoperative 3 months consultation

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided